CLINICAL TRIAL: NCT05537116
Title: Evaluation of an Interactive Mobile Phone-Based Brief Intervention to Reduce Substance-Impaired Driving Among Emerging Adults
Brief Title: Evaluation of an Interactive Mobile Phone-Based Brief Intervention to Reduce Substance-Impaired Driving
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-012
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Driving Impaired

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to conditions using a random number generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Personalized Feedback (Experimental): Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback. Feedback will include the following elements: a personalized substance use profile and substance-impaired driving profile, information on social norms related to substance use and substance-impaired driving, personalized information on BAC (or level of impairment due to drug use) prior to driving, costs associated with a DUI citation in Kentucky, and information on combined drug and alcohol impaired driving risk (if endorsed).
  Interventions: Behavioral: Personalized feedback
- Personalized feedback and text messages (Experimental): Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
  Interventions: Behavioral: Personalized feedback and text messages
- Information only (Active Comparator): Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
  Interventions: Behavioral: Information Only

INTERVENTIONS:
Behavioral: Personalized feedback — Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback. Feedback will include the following elements: a personalized substance use profile and substance-impaired driving profile, information on social norms related to substance use and substance-impaired driving, personalized information on BAC (or level of impairment due to drug use) prior to driving, costs associated with a DUI citation in Kentucky, and information on combined drug and alcohol impaired driving risk (if endorsed).
  Arms: Personalized Feedback
Behavioral: Personalized feedback and text messages — Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
  Arms: Personalized feedback and text messages
Behavioral: Information Only — Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
  Arms: Information only

SUMMARY:
Substance-Impaired Driving among emerging adults remains a significant public health concern and may be the single riskiest substance-related outcome among young adults. Brief Interventions (BIs) have been shown to reduce alcohol-impaired driving among this age group, but are not often implemented - despite their demonstrated efficacy - because it is not economically feasible to deliver in-person BIs to all emerging adult substance users. The present study will be the first to examine whether a text-messaging-based cannabis-impaired driving BI significantly decreases cannabis-impaired driving among emerging adult cannabis users compared to an informational control. Participants will be 240 emerging adults who endorse driving after cannabis use (or combined alcohol and cannabis use) at least three times in the past 3 months. After completing baseline measures, participants will be randomly assigned to receive either: a) substance use information, b) a substance-impaired driving personalized feedback intervention, or c) a substance-impaired driving personalized feedback intervention plus interactive text messages. Participants will complete outcome measures 3 and 6 months post-intervention. Repeated measures mixed modeling analyses will be used to determine whether the intervention significantly reduces substance-impaired driving over time. The project has two specific aims: 1) to evaluate a text based cannabis-impaired driving intervention in a randomized clinical trial, and 2) to determine whether the use of interactive text-messages sustains intervention effects over time.

DETAILED DESCRIPTION:
Rates of substance-impaired driving remain especially high among emerging adults, and substance-related traffic accidents remain the leading cause of substance-related death in this age group. Although rates of alcohol-impaired driving (AI-driving) among emerging adults have begun to decrease, rates of driving after cannabis use (DACU) continue to rise. In addition, many emerging adults report simultaneous use of alcohol and cannabis, a behavior that has been shown to increase the odds of substance-impaired driving and results in substantially greater fatal crash risk. Brief Interventions (BIs) have been shown to decrease substance use and related problems.6 BIs attempt to identify and correct faulty normative beliefs and highlight personal consequences of substance use (such as driving after substance use). BIs typically consist of one or two individual therapeutic meetings delivered in motivational interviewing (MI) style and include personalized feedback (based on a series of questionnaires completed by the participant prior to their BI session). One reason why BIs have not been widely implemented- despite their demonstrated efficacy - is that it is not economically feasible for universities and community agencies to hire and train staff to deliver in-person BIs to all substance users, and very few emerging adults seek out substance prevention or treatment services available on campus or in the surrounding community. Innovative ways of delivering BIs to this at-risk population, in a manner that is both effective and economically feasible, need to be developed. Text messaging represents a particularly advantageous way to provide BIs as they can be highly personalized to the individual and allows for engagement and interaction between the interventionist and participant. Research indicates that emerging adults prefer text messages to telephone calls and emails and rate this medium positively. Given the high prevalence and fatal consequences of substance-impaired driving, highly accessible intervention approaches are imperative for reducing this extremely risky behavior.

In the past few years, a number of interventions using text-messaging to target substance use and problems have been developed and evaluated with reviews and meta-analyses suggesting that the majority of these interventions result in improved outcomes and warrant further large scale studies. Most of these interventions target overall substance use and problems and do not focus on specific risk behaviors, such as substance-impaired driving. We have developed and evaluated a mobile-based BI focused specifically on decreasing AI-driving among college students in a pilot trial. This study indicated that a brief, mobile-based AI-driving intervention including MI text messaging resulted in significantly greater reductions in AI-driving at the 3-month follow-up, compared to alcohol information alone. We modified the intervention to focus on driving after cannabis use and found that the intervention resulted in significantly greater increases in perceived dangerousness of DACU and significantly greater decreases in DACU compared to to an informational control condition. Importantly, several recent studies have demonstrated greater effectiveness of interventions that include personal contact vs. those that are fully automated. The present study provides an important bridge between in-person therapist delivered interventions and fully automated interventions by utilizing interactive text messaging with participants in order to enhance retention of intervention elements and provide tailored, individualized interaction. It is imperative to directly test whether the use of interactive text-messages decreases substance-impaired driving significantly more than personalized feedback alone.

The proposed study will extend promising pilot results by: (a) increasing power by recruiting 240 emerging adults reporting recent driving after cannabis use (DACU), (b) including a 6-month follow-up to determine whether intervention effects persist over time, (c) examining mediators of intervention outcomes (e.g., changes in cannabis-related cognitions), and (d) providing additional intervention content focused on decreasing driving after combined use of alcohol and cannabis. The overarching goal is to use mobile technology to reduce driving after substance use among emerging adult cannabis users.

We will conduct a 3-group trial with 240 emerging adults (ages 18-25; project 50% female; 20% minority) recruited from a community in the Southeastern United States.

Group 1: substance impaired driving personalized feedback Group 2: substance impaired driving personalized feedback and Motivational Interviewing (MI) interactive text messages Group 3: substance use information (control) Aim 1: Evaluate a text based substance-impaired driving intervention in a Randomized Clinical Trial.

Hypothesis 1: Group 2 will report greater reductions in driving after cannabis use and driving after simultaneous alcohol and cannabis use 3- and 6-months post-intervention.

Aim 2: Evaluate mechanisms of intervention response. Hypothesis 1: Cognitive factors (e.g., changes in perceptions of dangerousness and consequences, peer norms, cannabis expectancies) will mediate intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to speak, read, and write in English
* Reports driving after using cannabis prior to driving at least three times in the past three months
* Reports having access to a motor vehicle, a valid driver's license, and plans to drive a vehicle in the next 6 months
* Reports access to a cell phone and willingness to read intervention material and exchange 3 texts post intervention with the study administrator
* Reports a valid email address

Exclusion Criteria:

* Currently in treatment for substance use

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Driving after cannabis use | 3 and 6 months post-intervention
  Number of times driving after cannabis use in the past 3 months

SECONDARY OUTCOMES:
Driving after combined alcohol and cannabis use | 3 and 6 months post-intervention
  Number of times driving after combined use of alcohol and cannabis in the past 3 months

OTHER OUTCOMES:
Peer norms | 3 and 6 months post-intervention
  Perceived peer norms will be assessed by asking participants to indicate "How much do you think a typical college student approves of driving a car after using marijuana?" on a 7-point Likert scale from 1 (strongly disapprove) to 7 (strongly approve).
Perceived dangerousness | 3 and 6 months post-intervention
  Perceived dangerousness related to DACU will be assessed by asking participants to indicate, "How dangerous do you believe it is to drive after marijuana use?" on a 4-point Likert scale from 1 (Not at all dangerous) to 4 (Very dangerous).
Perceived consequences | 3 and 6 months post-intervention
  Perceived consequences related to DACU will be assessed by asking participants to indicate their perceived likelihood of being stopped by the police, being drug tested, being arrested, and having an accident on a 4-point Likert scale from 1 (Not very likely) to 4 (very likely).
Cannabis Expectancies | 3 and 6 months post-intervention
  Cannabis expectancies will be assessed using the Marijuana Expectancies Questionnaire-Brief. Scores range from 6-30 with higher scores representing higher levels of positive and negative expectancies

CONTACTS AND LOCATIONS:
Overall Officials: Jenni Teeters, PhD, Principal Investigator — Western Kentucky University
Locations (1):
- Kelly Thompson Hall, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will consist of self-reported data from survey questionnaires and qualitative data from text-messaging sessions. Preliminary data will be shared via a presentation at a national conference in the second and third years of the project. After all data is collected, a manuscript detailing findings from the study will be submitted for peer-review and de-identified data will be submitted to the NIDA data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After all data is collected, a manuscript detailing findings from the study will be submitted for peer-review and de-identified data will be submitted to the NIDA data archive.